CLINICAL TRIAL: NCT06104748
Title: A Cohort of Maternal Vascular Malperfusion-related FGR (CoMVMFGR)
Status: Recruiting | Type: Observational
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Principal Investigator, Luming Sun, Professor, Shanghai First Maternity and Infant Hospital
Other Study IDs: ShanghaiFMIH-FMU6
Record Dates: First submitted 2023-10-16; First posted 2023-10-27 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: MVM-FGR
Keywords: FGR; maternal vascular malperfusion; Doppler; placenta; etiologies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Maternal serum and plasma samples will be used for omics analysis, amniotic fluid will underwent genetic testing (including karyotyping, chromosomal microarray analysis and exome sequencing), and/or infection testing. Placenta will perform pathological testing after delivery.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Based on a precise diagnostic standard process, through a multicenter study, we will establish a cohort focusing on placenta-mediated fetal growth restriction (FGR). Long-term follow-up will be conducted to seek predictive indicators for short-term and long-term adverse outcomes of maternal vascular malperfusion-related FGR (MVM-FGR).

DETAILED DESCRIPTION:
Fetal Growth Restriction (FGR) denotes the inability of fetal growth to attain its inherent genetic potential due to diverse pathological influences. It stands as a significant determinant of morbidity and mortality during the perinatal phase, intricately linked with adverse long-term consequences. The etiology of FGR is complex, involving maternal, placental/umbilical, and fetal factors. Among these, maternal vascular malperfusion-related FGR (MVM-FGR) emerges as the prevalent subtype, which is considered to have potential for early intervention and prevention.

To address this, we will establish a cohort dedicated to MVM-FGR, guided by a stringent diagnostic standard process tailored for FGR. Our objective is to compile a comprehensive dataset of singleton pregnancies diagnosed with MVM-FGR cases through multicenter collaboration. The definition of FGR aligns with the FIGO consensus criteria. We conduct thorough prenatal screenings for fetal factors, including genetic abnormalities, infections, and structural anomalies, subsequently enrolling MVM-FGR cases into our cohort.

Techniques including Doppler ultrasound, magnetic resonance imaging (MRI), and electronic fetal heart monitoring will be employed to assess fetal conditions. Follow-up continues until the child reaches the age of two years postpartum. Pathological examination of the placenta is performed after delivery, with additional placental genetic testing if necessary.

ELIGIBILITY:
Inclusion Criteria:

1.Singleton pregnancy 2. diagnosed as FGR according the delphi consensus:

1. Early-onset FGR(<32 weeks) Estimated fetal weight (EFW) or abdominal circumference (AC) < 3rd; or EFW or AC < 10th, combined with abnormal doppler, including uterine artery pulsatility index(UtA PI) >95th percentile, umbilical artery pulsatility index(UA PI) >95th percentile； or umbilical artery absent end-diastolic flow (UA-AEDF) or umbilical artery reversed end-diastolic flow(UA-REDF).
2. Late-onset FGR(≥32 weeks) Estimated fetal weight (EFW) or abdominal circumference (AC) < 3rd; or >2 of the following 3 criteria:

   * EFW or AC <10th percentile
   * EFW or AC crossing percentiles>2 quartiles on growth percentiles
   * CPR <5th percentile or UA-Pl>95th percentile 3.provision of signed written informed consent.

Exclusion Criteria:

* Fetus with definitive genetic disorders related to FGR, fetus with confirmed intrauterine infection (CMV, syphilis and etc.), fetus with structural anomalies
* Incomplete information or absence of informed consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women
Study Population: severe FGR singletons
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
short-term and long-term outcomes associated with MVM-FGR | during the pregnancy, up to an average gestational age of 40 weeks
  Exploration of short-term and long-term outcomes associated with MVM-FGR, encompassing intrauterine fetal demise, neonatal mortality, and severe neonatal morbidity.
predictive model for adverse outcomes | death during the pregnancy (average gestational age of 40 weeks), or death in 28 days after birth
  Development of a predictive model for adverse outcomes of MVM-FGR through the integration of maternal and fetal indicators

SECONDARY OUTCOMES:
Distribution of genetic etiologies of FGR | the day at birth
  Distribution of genetic etiologies of FGR under the standard assessment process.
Severe maternal complications | pregnancy-born after 28 days
  Severe maternal complications in MVM-FGR cohort

CONTACTS AND LOCATIONS:
Overall Officials: Luming Sun, Doctor, Principal Investigator — Department of Fetal Medicine, Shanghai First Maternity and Infant Hospital
Locations (1):
- Shanghai First Maternity and Infant Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided